CLINICAL TRIAL: NCT01512563
Title: Clinical Trial Comparing Patency and Safety of the Paclitaxel Eluting Covered Metallic Biliary Stent(Niti-S Mira-Cover Biliary Stent ) to the Common Covered Metallic Biliary Stent(Niti-S Biliary Stent)
Brief Title: Patency and Safety of the Drug Eluting Covered Biliary Stent Comparing to the Common Covered Biliary Stent
Acronym: MIRA-cover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MIRA-cover
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2012-01

CONDITIONS: Biliary Stricture; Malignant Neoplasms
Keywords: paclitaxel; drug eluting stent
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel ElutingCovered Metal Stent (Experimental)
  Interventions: Device: Biliary stent
- Covered Metal Stent (Active Comparator)
  Interventions: Device: Biliary stent

INTERVENTIONS:
Device: Biliary stent — palliative treatment for malignant patients
  Other Names: Niti-S Mira-Cover Biliary Stent; Niti-S Biliary Stent

SUMMARY:
Paclitaxel covered metal biliary stent extents their patency rate comparing to the Common Covered Metallic Biliary Stent.

DETAILED DESCRIPTION:
Paclitaxel covered metal biliary stent(Mira-Cover Biliary Stent) extents their patency rate comparing to the Common Covered Metallic Biliary Stent(Niti-S Biliary Stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is inoperable and/or unresectable cases of pancreatic cancer and/or biliary cancer with mid or distal CBD invasion
* Among patient of a.,Patient who previously had surgical biliary drainage of plastic stent have eligibility

Exclusion Criteria:

* Patient who have life expectancy under 3 months
* Patient who have severe metastasis of Liver or whole body
* Patient who previously had surgical biliary drainage

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Accumulative Patency Rate | 6 month

SECONDARY OUTCOMES:
Accumulative Survival Rate | 6 months
Complications | 6 months
Possibility of Other Treatment after Obstruction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Lee, Ph.D, Study Chair — Kangnam Severance Hospital; Ho Gak Kim, Principal Investigator — Catholic University of Daegu School of Medicine; Sang Heum Park, Principal Investigator — Soon Chun Hyang University
Locations (3):
- South Korea (3):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Catholic University of Daegu School of Medicine, Daegu
  - Kangnam Severance Hospital, Seoul